CLINICAL TRIAL: NCT05666050
Title: Effectiveness of Interactive Mobile Health Intervention (IMHI) to Improve Neonatal Care Practice Among Postpartum Women in Dessie and Kombolcha Town Zones, North East Ethiopia: Behavioral Cluster Randomized Control Trial
Brief Title: Mobile Health Intervention to Improve Neonatal Care Practice
Acronym: NCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wollo University (Other)
Collaborators: Jimma University (Other)
Responsible Party: Principal Investigator, Niguss Cherie, Assistant professor, Wollo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JUIH/IRB/230/22
Record Dates: First submitted 2022-12-05; First posted 2022-12-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Care
Keywords: Neonatal care, Dessie, Kombolcha, Ethiopia

STUDY DESIGN:
Intervention Model Description: Pregnant women with 26-28 weeks of gestation(based on world health organization eligibility criteria) will be recruited and baseline data will be collected at selected clusters. Women who will provide informed consent will be asked to complete a post-consent eligibility assessment including access to a mobile phone, and willingness to receive health messages on their mobile phone. Women who meet these eligibility criteria will be enrolled in the study and administered the baseline interview. Intervention will be started among randomly selected clustered pregnant women at 30 weeks of gestation and continued up to 6 weeks of post partum period for 4 months. Three intervention worker female nurses/midwifes will be recruited and trained to do the intervention based on the protocol After this end line data will be collected from both intervention and control group.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be masked about which group is intervention and control to avoid bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive mobile health intervention sending message service(SMS)
  Interventions: Behavioral: Mobile health intervention
- Control group (No Intervention): The control group will receive the existed current health delivery approach, no mobile health sending message service

INTERVENTIONS:
Behavioral: Mobile health intervention — Pregnant women with 26-28 weeks of gestation(based on world health organization eligibility criteria) will be recruited and baseline data will be collected at selected clusters. Women who will provide informed consent will be asked to complete a post-consent eligibility assessment including access to a mobile phone, and willingness to receive health messages on their mobile phone. Women who meet these eligibility criteria will be enrolled in the study and administered the baseline interview. Intervention will be started among randomly selected clustered pregnant women at 30 weeks of gestation and will be continued up to 6 weeks of post partum period for 4 months.
  Arms: Intervention group

SUMMARY:
Effectiveness of interactive mobile health intervention (IMHI) to improve neonatal care practice among postpartum women in Dessie and Kombolcha town zones, north east Ethiopia: behavioral cluster randomized control trial.

DETAILED DESCRIPTION:
The main aim of this study is to determine effectiveness of mobile health intervention to improve neonatal care practice among postpartum women in Dessie and Kombolcha town zones, North east Ethiopia. First participants will be grouped in to two arms based on randomization of clusters. The intervention arm will take the new intervention with existed health care practice and the control arm will take the existed current health care practice.

The intervention arm will receive sending message service (SMS) over a four month period (90 days pre-natal and 42 days post-partum) and the control arm will receive the existed health care practice. Participants in the intervention arm will receive mobile based health education and health communication messages as well as messages on neonatal care practice based on national maternal and child health care education and counseling guidelines. Participants in this study will be randomly assigned as intervention will receive sending message service from a trained professional; while participants assigned to control group will not receive phone based interventions but can contact their health care providers as routine health facility activity. Initially, study participants will receive one text message every two weeks with the frequency increasing to messages for 42 days following delivery.

Pregnant women with 26-28 weeks of gestation(based on world health organization eligibility criteria) will be recruited and baseline data will be collected at selected clusters. Women who will provide informed consent will be asked to complete a post-consent eligibility assessment including access to a mobile phone, and willingness to receive health messages on their mobile phone. Women who meet these eligibility criteria will be enrolled in the study and administered the baseline interview. Intervention will be started among randomly selected clustered pregnant women at 30 weeks of gestation and continued up to 6 weeks of post par-tum period for 4 months. Three intervention worker female nurses/midwifes will be recruited and trained to do the intervention based on the protocol After this end line data will be collected from both intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 26-28 weeks of gestation and have mobile phone access in the study area.

Exclusion Criteria:

* Pregnant women seriously ill and not able to respond.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 784 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Neonatal care practice among the intervention and control group will be measured by The minimum WHO 12 items will be used to produce composite index (score). | Two weeks after intervention the outcome will be measured.
  Principal component analysis will be done to create composite index (score) and respondents who will have scored above or equal to the mean/median value will be considered as having good neonatal care, while those who will score below the mean/median value were considered as poor neonatal care.

CONTACTS AND LOCATIONS:
Overall Officials: Niguss Cherie, Principal Investigator — Wollo Universirty
Locations (1):
- Dessie and Kombolcha, Dessie, South Wollo, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The data from the participants will be confidential.

REFERENCES:
- [Background] Cherie N, Abdulkerim M, Abegaz Z, Walle Baze G. Maternity continuum of care and its determinants among mothers who gave birth in Legambo district, South Wollo, northeast Ethiopia. Health Sci Rep. 2021 Nov 2;4(4):e409. doi: 10.1002/hsr2.409. eCollection 2021 Dec. PMID 34754945
- [Derived] Cherie N, Wordofa MA, Debelew GT. The effect of an interactive mobile health intervention to improve community-based essential neonatal care practices among postpartum women in northeast Ethiopia: a cluster randomized controlled trial. Int Health. 2025 Sep 3;17(5):820-835. doi: 10.1093/inthealth/ihae080. PMID 39789852